CLINICAL TRIAL: NCT04116398
Title: Pilot and Phase 2 Study of the Efficacy of a Treatment Protocol With Dexamethasone Implant Loading Dose in Patients With Diabetic Macular Edema
Brief Title: Pilot and Phase 2 Study of the Efficacy of a Treatment Protocol With Dexamethasone Implant Loading Dose in Patients With Diabetic Macular Edema (LOADEX)
Acronym: LOADEX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0588; 2019-003092-18 (EudraCT Number); 2024-514362-39-00 (EU CTIS Number)
Record Dates: First submitted 2019-09-16; First posted 2019-10-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Macular Edema
Keywords: dexamethasone,; loading dose,; diabetic macular edema; pseudophakic
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ozurdex®, 700µg dexamethasone intravitreal injection (Experimental): Intravitreal injection of dexamethasone (Ozurdex®)
  Interventions: Drug: Dexamethasone with 2 loading doses followed by PRN regimen.

INTERVENTIONS:
Drug: Dexamethasone with 2 loading doses followed by PRN regimen. — * Loading dose with 2 systematic intravitreal injections (IVI) of ozurdex at the baseline and 12 weeks.Followed by a PRN regimen with strict retreatment criteria (already used and published in the Prediamex study, Bellocq,Kodjikian et al Ophthalmology Retina 2017)
  * Retreatment criteria: Reduction in VA ≥ 5 ETDRS Letters; and/or CSMT ≥ 275 microns by OCT-Cirrus® or ≥ 285 microns by OCT Spectralis®/Topcon; and/or increase of CSMT > 50 microns; and/or onset of recurrent retinal cysts; and/or residual edema considered by the practitioner to be clinically significant.
  * Minimal time limit between two IVI : 12 weeks
  * Visits: monthly during 1 year (to check efficacy and safety) and then for the 2nd-year only at Month18 (M18) and Month 24 (M24)

SUMMARY:
Nowadays, steroids and anti-VEGF are the first line treatment for diabetic macular edema. Ozurdex is the most frequently used steroid and has label for both first and second line treatment. Ozurdex treatment paradigm for patients with diabetic macular edema is to inject patient only in case of huge recurrence. The risk of this scheme is a progressive loss of vision due to photoreceptors loss. A more pro-active regimen, as it already exists for anti-VEGF treatment, would allow a better patient management. A new treatment paradigm consisting in a loading dose of 2 injections within 12 weeks, followed by a PRN (Pro Re Nata) regimen with strict retreatment criteria and minimal time limit of 12 weeks between two injections should result in a better visual acuity gain and a limited augmentation of the number of injections (which will remain lower than the number observed for anti-VEGF treatment).

The investigators have therefore chosen a pilot study to investigate the impact on efficacy and on the number of intravitreal injections (IVI) of such a scheme.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 40 years old
* Patients with a significant DME : Macular thickening secondary to DME involving the center of the fovea, as measured by SD-OCT, with Central Subfield Thickness (CST) ≥ 285 μm measured on Spectralis/topcon or ≥ 275 μm, as measured on Cirrus, at screening and VA between 20/32 and 20/320 (between 23 and 78 letters ETDRS) using the ETDRS protocol at the initial testing distance of 4 meters at inclusion
* Patient for which a dexamethasone implant is chosen
* 100% naive eyes (no history of steroids or anti-VEGF)
* Pseudophakic for at least 3 months
* HBA1c < 10%
* Blood pressure < 160/95
* Patient who give voluntary signed informed consent
* Patient affiliated with the French universal health care system or similar
* Patient able to participated in all visits and medical examinations during the study
* If both eyes have to be treated, only one eye will be included : the eye with the lowest visual acuity at the baseline

Exclusion Criteria:

* Aphatic eye without posterior lens capsule.
* Study eye with implant anterior chamber of the eye or intraocular implant with iris fixated or transsclerally or ruptured posterior lens capsule.
* Study eye with lens implant ARTISAN®
* Ocular or periocular infection active or suspected in the study eye including most viral diseases of the cornea and conjunctiva, epithelial keratitis active Herpes simplex (dendritic keratitis), vaccinia, chickenpox, mycobacterial infections and mycoses
* At inclusion, delay after cataract surgery < 3 months in the study eye
* Delay after last session of panretineal Photocoagulation laser < 1 month in the study eye
* Delay after last focal laser session of the posterior pole < 1 month in the study eye
* Vitreomacular traction syndrome, associated ERM in the study eye
* History of macular grid laser in the study eye
* Focal laser only if the scars are located within 750 microns of the center (1/2 Papillary Diameter) in the study eye
* Ischemic maculopathy (increase of more than 2 times the surface of the central avascular zone)
* Proliferative diabetic Retinopathy in the study eye
* Hypertension or Open Angle Glaucoma (OAG) treated by dual therapy eye drops or more
* Patients with a systemic pathology that could interfere in the evolution of the Diabetic Macular Edema and treated by with immunosuppressive drugs, systemic steroids, anti-aldosterone or systemic anti-VEGF.
* Patients with systemic treatment with a toxic effect on the lens, retina or optic nerve: deferoxime, chloroquine / hydroxychloroquine, tamoxifen, phenothiazines and ethambutol; in progress or within 6 months of inclusion
* Hypersensitivity to the active substance or to any of the excipients and to anesthetic or hypotonizing eye drops
* History of any pathology, metabolic disease, or any serious suspicion of disease at clinical or laboratory examination that contraindicates the use of the intra-retinal dexamethasone implant, could affect the interpretation of the results of the study or cause significant risks of complication for the subject
* Infectious conjunctivitis and/or active or suspected appendix infection
* Any eye condition or condition that the investigator believes may require intraocular surgery within 12 months
* Eye contralateral that studied with visual acuity < 23 letters
* Pregnant and breastfeeding woman
* Female of reproductive age, sexually active, who does not want to commit to using adequate and highly effective contraception during the study and up to 6 months after the last administration of the study treatment:

  * Combined hormonal contraception (containing estrogens and progestins) aimed at inhibiting ovulation (oral, intravaginal or transdermal);
  * Hormonal contraception containing only a progestin intended to inhibit ovulation (oral, injectable or implantable);
  * Intrauterine device (IUD);
  * Intrauterine Hormone Release System (IUS);
  * Ovariectomy with hysterectomy, bilateral tubal obstruction or total hysterectomy for at least 6 weeks before inclusion (for women included) or vasectomy for at least 6 months before inclusion (for partners of a patient included);
  * Sexual abstinence. A woman will be considered to be of childbearing age from her first period and until the menopause, unless she is sterile or has had an oophorectomy type surgery with hysterectomy, bilateral tubal obstruction or hysterectomy total at least 6 weeks before inclusion. A post-menopausal state is defined as the absence of spontaneous menstruation (that is to say without any other medical treatment, in particular of the hormonal contraceptive type or hormone replacement therapy) for 12 months
* Major patient protected under the terms of the law (Public Health Code)
* Patient's ongoing participation in another interventional clinical trial (study eye and/or untreated eye)
* Follow-up impossible for 24 months, the judgment of the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum BCVA (Best Corrected Visual Acuity) change (best improvement) from baseline (during one year of treatment) | 52 weeks
  Best Corrected Visual Acuity (BCVA) is measured on the ETDRS scale at an initial distance of 4 meters.

SECONDARY OUTCOMES:
The time required to obtain the best BCVA | 52 weeks
  average, standard deviation, median, minimum and maximum
The number of injections required to obtain the best BCVA | 52 weeks
  average, standard deviation, median, minimum and maximum
the maximum best corrected visual acuity (BCVA) change (best improvement) measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) scale | between the baseline and 1,5 years and between the baseline and 2 years
  Best Corrected Visual Acuity (BCVA) is measured on the ETDRS scale at an initial distance of 4 meters.
values of Visual Acuity (VA) at each visit | all visits during 2 years
Area under the curve (AUC) of VA | between the baseline and 52 weeks and between the baseline and 2 years
  AUC calculated with the values of VA at each visit
Description of Visual acuity (VA) | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
  categorized change of VA (>=+15 ; +10 -> +15 ; +5 -> +10 ; -5 -> +5 (stable) ; -5 -> -10 ; -10 -> -15 ; > -15)
Number of IVI | 1 year
Number of IVI | 2 years
OCT parameters: Central Subfield Mean Thickness (CSMT) | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
  average, standard deviation, median, minimum and maximum
OCT parameters: Central Fovea Thickness | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
  average, standard deviation, median, minimum and maximum
OCT parameters : presence of interruptions of the ellipsoid line | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
OCT parameters : presence of continuous external limiting membrane | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the which obtained the BCVA
OCT parameters : presence of disorganization of the internal retinal layers | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
OCT parameters : presence of intraretinal cysts | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
OCT parameters : presence of vitreomacular traction | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtain the BCVA
OCT parameters : presence of epiretinal membrane | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
OCT parameters : presence of macular exudates | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
OCT parameters : persistance of foveolar depression | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 years, 2 years and the visit which obtained the BCVA
OCT parameters : presence of intraretinal fluid | at each visit
Proportion of patients with macular edema resolution | at 1 year
  A macular edema resolution will be defined as absence of intraretinal fluid for at least 6 months after the last
Proportion of patients with macular edema resolution | at 2 years
  A macular edema resolution will be defined as absence of intraretinal fluid for at least 6 months after the last
Retinopathy parameters : presence of intraretinal or subretinal macular hemorrhage | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  on stereoscopic 7-field color fundus photographs
Retinopathy parameters: presence of microaneurisms | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  on stereoscopic 7-field color fundus photographs
Retinopathy parameters : presence of macular exudates | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  on stereoscopic 7-field color fundus photographs
Severity evolution (improvement, no change, worsening) of diabetic retinopathy graded by 2 evaluators on stereoscopic 7-field color fundus photographs | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  Using the Stadification Diabetic Retinopathy Severity Scale (DRSS), 5 levels: No apparent retinopathy, Mild Non Proliferative Diabetic Retinopathy (NPDR), Moderate NPDR,severe NDPR and Proliferative Diabetic Retinopathy (PDR)
Quantitative OCT-angiography analysis : the size of non-perfusion zones | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  The mean (and standard deviation) the median (minimum-maximum) of the size of non-perfusion
Quantitative OCT-angiography analysis : the size of central avascular zones | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  The mean (and standard deviation) the median (minimum-maximum) of the size of central avascular zones compared with baseline
Qualitative OCT-angiography analysis : presence of macular ischemia | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  the number of macular ischemia
Qualitative OCT-angiography analysis : Evolution of macular ischemia compared to the baseline | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  Types of evolution compared to baseline : appearance / disappearance / stability of the macular ischemia.
Qualitative OCT-angiography analysis : presence of preretineal neovessels | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  the number of preretineal neovessels,
Qualitative OCT-angiography analysis : evolution of preretineal neovessels compared to the baseline | Baseline, 12 weeks, 24 weeks,36 weeks,52 weeks, 1.5 year and 2 years
  Types of evolution : appearance / disappearance / stability.
Biomicroscopy: the number and the percentage by categories of the condition of the implant | all visits during 2 years
  conditions : clear, opacified , integrity, open, performed capsulotomy
Biomicroscopy: presence of the state of the posterior capsule | all visits during 2 years
  absence or presence of the posterior capsule
Variation of the intraocular pressure | all visits during 2 years
proportion of patients using hypotonic eye treatment | all visits during 2 years
Number of adverse events | all visits during 2 years
  All adverse events will be coded using the Meddra system organ class and cases of patients stopping or switching drugs will be described (causes, new drugs,..)
Level of discomfort felt by the patient | all visits during 1 year
  Discomfort felt by the patient measured by a visual analog scale (EVA between 0 and 10 (0 = no discomfort))

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - APHP - Hôpital Avicenne, Bobigny
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - Centre Rétine Gallien, Bordeaux
  - Hôpital Intercommunal de Créteil, Créteil
  - CHU Dijon, Dijon
  - CHRU Lille - Hôpital Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hospices Civils de Lyon - Hopital de la Croix Rousse, Lyon
  - Centre Monticelli Paradis d'ophtalmologie, Marseille
  - APHM - Hôpital Nord, Marseille
  - Clinique Juge, Marseille
  - APHP - Hôpital Lariboisière, Paris
  - Centre Hospitalier National d'Ophtalmologie des XV XX, Paris
  - CHU de Poitiers - La miletrie, Poitiers
  - Clinique Mathilde, Rouen
  - CHU Toulouse - Hôpital Pierre Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided